CLINICAL TRIAL: NCT06490822
Title: The Skin as a Window to the Central Nervous System in Frontotempolar Lombar Degeneration
Acronym: PROTEINOSKIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC23_0575
Record Dates: First submitted 2024-06-25; First posted 2024-07-08 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Frontotemporal Lobar Degeneration
Keywords: FTLD; tau; TDP43; skin biopsy
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Pick Disease of the Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Other): A single 3 mm-diameter punch skin biopsy will be obtained from FTLD patients and healthy volunteers at the C8 paravertebral under local anesthesia to analyze cutaneous innervation
  Interventions: Procedure: Skin biopsy

INTERVENTIONS:
Procedure: Skin biopsy — A single 3 mm-diameter punch skin biopsy will be obtained from FTLD patients and healthy volunteers at the C8 paravertebral under local anesthesia to analyze cutaneous innervation

SUMMARY:
Frontotemporal lobar degeneration (FTLD) is a clinically heterogeneous syndrome, characterized by progressive decline in behaviour and/or language. From a pathological standpoint, like the great majority of neurodegenerative disorders, FTLD are proteinopathies, which are characterized by the presence of specific protein deposits in the Central Nervous System (CNS). Accordingly, the two main deposits observed in FTLD are either made of Tau or transactive response DNA binding protein 43 (TDP-43).

In pathological conditions such as FTLD, both proteins are aggregated and hyperphosphorylated.

It is now well established that the pathological process in some proteinopathies such as synucleinopathies (of which Parkinson's disease is the main representative) is not limited to the brain but also widespread throughout the peripheral autonomic networks, including the autonomic innervation of the skin. In this context, many independent studies have shown that the pathological process in PD could be detected using routine punch skin biopsies opening the way for the development of original histopathological markers of the disease.

Our hypothesis is that such a scenario could also occur in FTLDs and that the detection of the pathological tau or TDP-43 protein in the skin could help in diagnosing FTLD. This is especially relevant as, despite the recent progress in genetics, neurobiology and neuroimaging, there are no available biomarkers for FTLD.

DETAILED DESCRIPTION:
Participant with Frontotemporal Lobar degeneration equally distributed into behavioral variant of frontotemporal dementia (bvFTD), language variant with primary progressive aphasia (PPA) and motor presentations with atypical parkinsonian disorders (corticobasal degeneration-CBD and progressive supranuclear palsy-PSP) and motoneuron disorder (amyotrophic lateral sclerosis -ALS) will be included at Nantes University Hospital during a period of 24 months.

Healthy volunteers will be included as comparative group. A skin biopsy and venous blood samples will be collected for all participants.

ELIGIBILITY:
Inclusion Criteria (patients):

* Adressed or followed at memory clinic or ALS expert center at Nantes university hospital.
* Aged 50-75 years
* Fulfilling current diagnosis criteria for one of the disorder: vcfFTD, non-Alzheimer PPA (semantic or non fluent), DCB or PSP,ALS
* MMSE ≥ 18
* Membership of social security scheme

Inclusion Criteria (healthy volunteers):

* No history of neurological disease, diabetes, or alteration/damage of peripheral nervous system
* Aged 50-75 years Paired to at least one patient on age (less or more 5 years)
* MOCA ≥ 26
* Membership of social security scheme

Non inclusion Criteria (Patients and healthy volunteers):

* Concomitting conditions affecting the peripheral nervous system such as but not limited to diabetes, renal failure, thyroid disorder, vitamin B12 deficiency, acute and chronic inflammatory diseases HIV, syphilis
* Know allergy to local anesthetic
* Known coagulopathy
* Pregnant women or breastfeeding women
* Person under court protection sous sauvegarde de justice
* Person under guardianship
* Inability to sign an informed consent

Non inclusion criteria (Patients) • Patient with neurological disease other than FTLD

Non inclusion criteria (Healthy volunteers) :

• Evidence of neurological disorder at the inclusion including but not limted to FTLD, Parkinson disease, Alzheimer disease, lewy body dementia, Huntington disease, systemic lupus erythematosus multiple sclerosis; learning disabilities, mental retardation, severe hypoxic brain injuries, brain trauma with permanent cognitive impairments.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Amount of TDP 43 | Day of inclusion
  assessed by Western blot and qPCR to determine level of expression of TDP-43 in the skin
Amount of Tau assessed by Western blot and qPCR | Day of inclusion
  assessed by Western blot and qPCR to determine level of expression of Tau in the skin

SECONDARY OUTCOMES:
Amount of Tau phosphorylation | Day of inclusion
  phospho-tau/tau ratio in the skin will be measured by Western blot
Amount of TDP 43 phosphorylation | Day of inclusion
  phospho-TDP-43 /TDP43 ratio in the skin will be measured by Western blot
Neuropsychological characterization | day of inclusion for patients vFTD, PPA and corticobasal degeneration-CBD and progressive supranuclear palsy-PSP within 12 months of inclusion for patients ALS
  During their follow-up FTLD patients underwent a complete neuropsycological assessment define as:
  * mini-mental state examination (MMSE)
  * the 16-item Free Recall/Indicated Recall test (RL/RI-16 items)
  * Rey figure and recall
  * Trail Making Test (TMT A & B)
  * Wechsler Adult Intelligence Scale
  * Literal (letter P) and categorical (animals) fluency
  * Rapid Frontal Efficiency Battery (BREF)
  * Wisconsin Card Sorting Test (WCST)
  * Zoo test of Behavioural Assessment of the Dysexecutive Syndrome (BADS)
  * Stroop test - 4 boards
  * Oral image naming test (DO 80)
  * Theory of mind (ToM-15)
  * ekman facial emotion recognition test
Behaviour profile | day of inclusion for patients vFTD, PPA and corticobasal degeneration-CBD and progressive supranuclear palsy-PSP within 12 months of inclusion for patients ALS
  The 10-items scale Daphne will be used to explore disinhibition (4 items), apathy(1 item), perseveration (1 item), hyperorality (2items), personal neglect (1 item) and loss of empathy (1 item)
FTLD mutation | before inclusion
  Mutation carrier patient will be identified among participant (not all the participant) who had a genetic screening had neen carried out during their follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France